CLINICAL TRIAL: NCT06114550
Title: Acute Effect of Resistance Training With Different Intensity on Circulating Levels of Neurotrophic Growth Factors and Homocysteine in Young Adults
Brief Title: Resistance Training on Growth Factors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Chongwen Zuo, Doctoral, Air Force Military Medical University, China
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: zuochongwen
Record Dates: First submitted 2023-10-24; First posted 2023-11-02 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Cognitive Function
Keywords: neurotrophic growth factors; IGF-1; BDNF; VEGF; Irisin; Hcy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity resistance training group (HIRT) (Experimental): All subjects were instructed to conduct HIRT consisted of 4-5 sets of 12 repetitions at 80%1RM, with 1-2 minutes rests between each set.
  Interventions: Other: High intensity resistance training
- low-intensity resistance training group (LIRT) (Experimental): All subjects were instructed to conduct LIRT consisted of 4-5 sets of 24 repetitions at 40%1RM, with same period) in random order.
  Interventions: Other: Low intensity resistance training

INTERVENTIONS:
Other: High intensity resistance training — The HIRT protocol comprised five exercises (bench press, barbell back squat, deadlift, seated leg flexion, and reverse arm curl) at 80% of 1RM, and 4-5 sets of 12 repetitions with 1-2 minutes of rest period between sets for approximately 60 minutes.
  Arms: High-intensity resistance training group (HIRT)
Other: Low intensity resistance training — For LIRT protocol, which performed same training exercises as HIRT. The repetitions in the LIRT protocol were assessed using the following equation: 80% of 1RM lifting load (kg) ×repetitions (HIRT)/40% of 1RM to volition fatigue, with 1-2 minutes of rest period between sets. Therefore, the LIRT protocol completed 4-5 sets of 24 repetitions at 40% of 1RM for a total of 60 minutes.
  Arms: low-intensity resistance training group (LIRT)

SUMMARY:
The goal of this clinial trial study is to explore the effect of high or low intensity resistance training (LIRT) under similar training volume on change in serum levels of BDNF, IGF-1, VEGF, irisin, and plasma Hcy in young adults.The main questions it aims to answer are:

1. Whether high and low intensity will increase the serum levels of BDNF, IGF-1, VEGF, irisin, and reduce plasma Hcy.
2. whether a greater magnitude of change would be suffer in low intensity group when compared to high intensity group, as an effect of greater physiological adaptation produced by more repetitions required to complete.

Participants will performe two different intensity resistance training (HIRT, at 80%1RM with 12 repetitions and 4-5 sets and LIRT, at 40%1RM with 24 repetitions and 4-5 sets).

Researchers will compare the training effects of two different training on these growth factors.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 to 30 years
* no experiencing musculoskeletal disorders or sports injuries
* had not participated any regular aerobic endurance or resistance training with in the previous half years
* no smoking habit or intake alcohol and other medication (e.g., steroid hormone)
* good general body condition without any chronic diseases (e.g., osteoarthritis, metabolic syndrome or arthritis)

Exclusion Criteria:

* experiencing musculoskeletal disorders or sports injuries in recent 1 month
* had regular resistance training exercise
* intake any supplementary(drug and hormone)

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-02-27 (Estimated); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-04-07 (Estimated)

PRIMARY OUTCOMES:
Rata of perceived exertion | "0 minutes" "60 minutes" "90 minutes"
  The rating of perceive exertion (RPE) questionnaire scale was applied to assess participants' subjective fatigue feeling throughout the training period.
Blood lactate | "0 minutes" "60 minutes" "90 minutes"
  serum blood lactate
BDNF | "0 minutes" "60 minutes" "90 minutes"
  regulators of neurogenesis
IGF-1 | "0 minutes" "60 minutes" "90 minutes"
  regulators of neurogenesis
VEGF | "0 minutes" "60 minutes" "90 minutes"
  regulators of neurogenesis
Irisin | "0 minutes" "60 minutes" "90 minutes"
  regulators of neurogenesis
Hcy | "0 minutes" "60 minutes" "90 minutes"
  homocysteine (Hcy) increase with age and resulted in cognitive function decline through greater oxidative stress and vascular dysfunction

SECONDARY OUTCOMES:
Reactive time | "0 minutes" "60 minutes" "90 minutes"
  Reaction time is the time it takes for the body to go from receiving a stimulus to responding to an action
Accuracy rate | "0 minutes" "60 minutes" "90 minutes"
  Accuracy refers to the correct degree of expression or description of a thing, which is used to reflect the correct answer to the thing

CONTACTS AND LOCATIONS:
Overall Officials: chongwen zuo, Doctoral, Principal Investigator — Air Force Medical Center of Chinese PLA

IPD SHARING:
Plan to Share IPD: Yes
The raw data supporting the conclusions of this article will be made available by the authors, without undue reservation, to any qualified researcher. First author should be contacted if someone wants to request the data from this study.
Supporting Information: SAP
Time Frame: When this study was published.
Access Criteria: Shall not be used for secondary analysis or repeated publication
URL: http://www.medresman.org.cn